CLINICAL TRIAL: NCT04807413
Title: Nitric Oxide During Cardiopulmonary Bypass in Adult Surgery: A Randomized Double Blinded Trial
Brief Title: Nitric Oxide During Cardiopulmonary Bypass in Adult Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0056-21
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-03

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm: The balloon will be opened to deliver nitric oxide at 40 ppm. (Experimental): Nitric oxide balloon will be connected to the CPB machine. Participants randomized to this group will receive 40 ppm nitric oxide through the pump.
  Interventions: Drug: Nitric Oxide
- Control Arm: The balloon will be closed and no nitric oxide will be delivered. (Active Comparator): Participants in this group will receive standard of care treatment. Participation in the trial will not affect surgery management in any way.
  Interventions: Other: standard of care treatment

INTERVENTIONS:
Drug: Nitric Oxide — The balloon will be opened to deliver nitric oxide at 40 ppm through the cardiopulmonary bypass machine
  Arms: Study Arm: The balloon will be opened to deliver nitric oxide at 40 ppm.
Other: standard of care treatment — standard of care treatment
  Arms: Control Arm: The balloon will be closed and no nitric oxide will be delivered.

SUMMARY:
Inhaled nitric oxide is a widely accepted standard of care for pulmonary hypertension, and has been studied in the context of cardiac surgery. CPB during cardiac surgery induces systemic inflammatory response and ischemic-reperfusion injury of many organs. Nitric oxide added to the bypass circuit may have anti-inflammatory effect and has shown the potential to ameliorate organs' injury .

There is evidence that the delivery of nitric oxide to the oxygenator gas flow during pediatric CPB is accompanied by a reduction in myocardial injury markers' levels in the postoperative period. In adults, NO supply to the CPB circuit during CABG exerted a cardioprotective effect and was associated with a lower level of inotropic support and cardio-specific blood markers .

To our knowledge, this is the first trial to assess whether artificial nitric oxide supplementation to the CPB-system reduces the incidence of hypoxemia after cardiac surgery.

DETAILED DESCRIPTION:
This prospective, single center, double blinded, interventional trial will be conducted at Rabin Medical Center Beilinson Hospital. Adult patients undergoing CABG and valve replacement/ repair surgeries will be eligible to participate.

All The participant will sign an informed consent prior to any procedures being done specifically for the purpose of the study, in the departmental ward on the day of surgery when they are not under the influence of sedatives and are not in pain. The study design and patient requirements will all be explained to the patient by the study investigator throughout the consent process. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. All consent forms will be IRB-approved. Each participant will receive a signed copy of the informed consent document for their record.

Treatment allocation will be performed by an independent investigator who will not be directly involved in the participants' treatment.

All other study investigators will be blinded to a group assignment. All study participants will be blinded to a treatment arm allocation. Upon consent, all study participants will be randomized in a 1:1 ratio to one of the two study arms.

Nitric oxide balloon will be connected to the CPB machine. Study Arm: The balloon will be opened to deliver nitric oxide at 40 ppm. Control Arm: The balloon will be closed and no nitric oxide will be delivered. Following randomization, all study participants will undergo the surgery according to standard clinical practice. In the surgery room all study participants will be connected to a standard anesthesia monitor and will be monitored according to standard clinical practice, which will include monitoring according to ASA standards, insertion of an arterial line and a CVP catheter.

Participation in the study will not affect the anesthetic, surgical and cardiopulmonary bypass management in any way. The anesthetic protocol administered to the study participant is at the attending anesthesiologists' discretion.

In addition to treatment arm allocation, all study participants will be monitored during surgery and followed-up throughout their duration of stay in the ICU and at the department ward.

Throughout the follow-up, study participants' blood tests and vital signs, as routinely monitored, will be collected and documented.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective CABG surgeries with CPB at Rabin Medical Center Beilinson hospital.
2. Patients undergoing valve replacement/repair surgeries with CPB at Rabin Medical Center Beilinson hospital.

Exclusion Criteria:

1. Patients requiring ECMO use preoperatively.
2. Patients requiring IABP use preoperatively.
3. Patients experiencing preoperative shock (defined as the need for ionotropic and/or vasopressor support).
4. Patients after solid organ transplant surgery.
5. Patients with LVAD.
6. Patients with ESRD requiring dialysis preoperatively.
7. Patients with a language barrier.
8. Patients unable to give informed consent.
9. Patients with heparin induced thrombocytopenia.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative hypoxemia | Within 24 hours postoperatively

SECONDARY OUTCOMES:
Incidence of Low cardiac output syndrome | Within 72 postoperatively
Use of drugs for hemodynamic support such as phenylephrine, noradrenaline | Within 72 postoperatively
Incidence of Acute Kidney Injury | Within 72 postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Eidelman, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center/Beilinson Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azem K, Novakovsky D, Krasulya B, Fein S, Iluz-Freundlich D, Uhanova J, Kornilov E, Eidelman LA, Kaptzon S, Gorfil D, Aravot D, Barac Y, Aranbitski R. Effect of nitric oxide delivery via cardiopulmonary bypass circuit on postoperative oxygenation in adults undergoing cardiac surgery (NOCARD trial): a randomised controlled trial. Eur J Anaesthesiol. 2024 Sep 1;41(9):677-686. doi: 10.1097/EJA.0000000000002022. Epub 2024 May 28. PMID 39037709